CLINICAL TRIAL: NCT02083510
Title: A Translational Study to Understand the Mechanism of Apolipoprotein CIII Reduction Via Colchicine
Brief Title: Apolipoprotein CIII Reduction Via Colchicine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Peter G. Schultz, PhD, Prinicpal Investigator, The Scripps Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-6293; 1UL1TR001114-01 (NIH)
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Hypertriglyceridemia; Gout; Pericarditis
Keywords: Colchicine; Hypertriglyceridemia; Apolipoprotein CIII
MeSH Terms: conditions — Hypertriglyceridemia; Gout; Pericarditis | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colchicine (Experimental): Patients will be enrolled with either gout/pericarditis or hypertriglyceridemia, have VAP and Apolipoprotein CIII levels at baseline, administer Colchicine for 6 weeks with reassessment of Apolipoprotein CIII and VAP.
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine
  Other Names: Colcrys

SUMMARY:
The aim of this trial will be to determine an effect-size for the administration of chronic low-dose colchicine in the reduction of serum levels of triglycerides (TG), very-low density lipoproteins (VLDL), and apolipoprotein CIII (apoCIII) in human subjects over a period of 4-6 weeks.

DETAILED DESCRIPTION:
The aim of this proposal will be to show, in a translational fashion, a relationship between colchicine and reduction of factors affecting triglyceride metabolism, especially apoCIII and VLDL levels. We envision colchicine as playing a role in identifying and elucidating a new mechanism for lowering TG levels, which may have a great impact on targeting patients who have not met non-HDL goals according to Adult Treatment Panel III (ATPIII guidelines) or at risk for hypertriglyceridemia-induced pancreatitis [11]. We will accomplish this by conducting a prospective cohort clinical trial of low-dose colchicine in hypertriglyceridemic patients to assess percent (%) reduction of apoCIII, VLDL, and TG. Secondary endpoints will be to observe the effects of colchicine on apoA, apoB, HDL, low-density lipoprotein (LDL), and total cholesterol (TC).

ELIGIBILITY:
Inclusion Criteria:

* Acute new-onset pericarditis or recurrent pericarditis (≥2 following criteria)

  * Sharp and pleuritic chest pain improved or relieved by sitting up and leaning forward
  * A pericardial friction rub
  * Electrocardiogram (EKG) findings of diffuse ST-segment elevations or PR depression
  * New or worsening pericardial effusion visualized on echocardiogram.

OR

•Acute gouty arthritis (according to the ACR; ≥1 of following criteria:

* Joint fluid containing urate crystals
* Tophus proved to contain urate crystals by chemical means
* Polarized light microscopy
* Presence of six of the following in the absence of crystal identification:
* >1 attack of acute arthritis
* Maximum inflammation developed in 1 day
* Monoarthritis attack
* Redness observed over joints
* 1st metatarsal joint painful or swollen
* Unilateral 1st metatarsal joint attack
* Unilateral tarsal joint attack
* Tophus (suspected)
* Hyperuricemia
* Asymmetric swelling within a joint visible on physical examination or radiography
* Subcortical cysts without erosions visible on radiography
* Monosodium urate monohydrate microcrystals in joint fluid during attack
* Joint fluid culture negative for organisms during attack.

If N < 10 after 3 weeks of trial initiation, then employ enrollment strategy #2

Enrollment strategy #2:

* History of hypertriglyceridemia (TG ≥ 150 mg/dL) AND
* Age ≥ 18 years old
* Capable of providing informed consent
* Capable of taking Colchicine 0.6-1.2 mg/day orally for 6 weeks
* Capable of providing a blood sample

Exclusion Criteria:

* Colchicine use < 8 weeks from baseline VAP panel
* Pregnant or female of child bearing age
* On corticosteroid therapy or corticosteroid use < 4 weeks from baseline VAP panel
* History of statin myopathy or hepatotoxicity
* History of colchicine intolerance or hypersensitivity
* Severe end-stage renal disease (eGFR ≤ 20 mL/min/1.73 m2) or requiring dialysis
* Hepatic Impairment (Child-Pugh class B or C)
* Myopericarditis (If TnI is elevated on presentation of acute pericarditis)
* Inflammatory Bowel Disease
* Tuberculous, neoplastic, or purulent pericarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Reduction in ApoCIII levels | 6 weeks
Reduction of triglycerides and very low density lipoprotein (VLDL) levels | 6 weeks

SECONDARY OUTCOMES:
Measurement of Apolipoprotein A and Apolipoprotein B via Vertical Auto Profile (VAP) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schultz, PhD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States